CLINICAL TRIAL: NCT03699462
Title: The Effect of Balanced Crystalloid Versus 5% Albumin on Endothelial Glycocalyx Degradation in Patients Undergoing Off-pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2018-0670
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Occlusive Disease(CAOD)
Keywords: Endothelial Glycocalyx (EG); 5% albumin; off-pump coronary artery bypass surgery (OPCAB)
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Intervention Model Description: Groups are divided into 2 groups; those receiving balanced crystalloid solution (Plasma solution-A injection, CJ Pharma, South Korea), and those receiving 5% albumin (Albumin 5% inj, Green cross, South Korea) during surgery
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: One researcher (Anesthesiologist) conducts randomized group assignment, and the researcher is not involved in other aspects of anesthesia and research.
  Therefore, other researchers, and all those involved in anesthesia, surgery, and postoperative management do not know the patient's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma A group (Active Comparator): The group receiving balanced crystalloid solution (Plasma solution-A injection, CJ Pharma, South Korea) during surgery
  Interventions: Drug: Plasma solution-A injection
- Albumin group (Experimental): The group receiving receiving 5% albumin (Albumin 5% inj, Green cross, South Korea) during surgery
  Interventions: Drug: 5% Albumin

INTERVENTIONS:
Drug: Plasma solution-A injection — The group receiving balanced crystalloid solution (Plasma solution-A injection, CJ Pharma, South Korea) during surgery
  Arms: Plasma A group
Drug: 5% Albumin — The group receiving 5% albumin (Albumin 5% inj, Green cross, South Korea) during surgery
  Arms: Albumin group

SUMMARY:
It is being revealed that the more severe the damage of the endothelial glycocalyx (EG) layer, the more likely it is that the prognosis of the patients is poor. For that reason, research is being actively conducted on methods for reducing damage and promoting recovery of the EG layer.The natural regeneration process of the EG layer is up to 7 days. Considering the fact that it is quiet slow, reducing the damage of EG layer is considered to be very important for improving the prognosis of patients undergoing surgery, but there is no clinically proven method.

One of the ways receiving attention to reduce damage of EG layer is to stabilize the layer through fluid therapy with albumin. The purpose of this study is to compare the protective effect of the EG layer according to the type of fluid (balanced crystalloid solution vs. 5% albumin) during surgery in patients undergoing off-pump coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years of age undergoing off-pump coronary artery bypass surgery

Exclusion Criteria:

* Emergency operation
* Minimally-invasive surgery (under one-lung ventilation)
* Chronic kidney disease (eGFR<30 ml/min/1.73m2) or Dialysis
* Acute kidney injury
* Infectious disease
* Preoperative steroid use
* Malignancy
* Reported allergic reaction to albumin preparations
* Patients who participated in other clinical studies that could affect prognosis
* Patients who have difficulty in reading the informed consent and voluntarily agreeing to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-10-17 (Actual); Study Completion 2020-10-17 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Syndecan-1 | Before induction of anesthesia (1-hour before the start of surgery)
  The investigators compare the protective effect of EG layer according to the type of fluid used during surgery in patients undergoing off-pump coronary artery bypass surgery. (Comparison of the plasma concentration of Syndecan-1 between the two groups.)
Plasma concentration of Syndecan-1 | At the time of returning the heart in place after coronary artery anastomoses (1~2 hour before the end of surgery)
  The investigators compare the protective effect of EG layer according to the type of fluid used during surgery in patients undergoing off-pump coronary artery bypass surgery. (Comparison of the plasma concentration of Syndecan-1 between the two groups.)
Plasma concentration of Syndecan-1 | At the time of sternum being closed (30min~1hr before the end of surgery)
  The investigators compare the protective effect of EG layer according to the type of fluid used during surgery in patients undergoing off-pump coronary artery bypass surgery. (Comparison of the plasma concentration of Syndecan-1 between the two groups.)

SECONDARY OUTCOMES:
Plasma concentration of Haparan sulfate | Before induction of anesthesia (1hr before the start of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Plasma concentration of Haparan sulfate | At the time of returning the heart in place after coronary artery anastomoses (1~2hr before the end of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Plasma concentration of Haparan sulfate | At the time of sternum being closed (30min~1hr before the end of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Plasma concentration of ANP | Before induction of anesthesia (1hr before the start of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Plasma concentration of ANP | At the time of returning the heart in place after coronary artery anastomoses (1~2hr before the end of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Plasma concentration of TNF-α/IL-6 | Before induction of anesthesia (1hr before the start of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Plasma concentration of TNF-α/IL-6 | At the time of sternum being closed (30min~1hr before the end of surgery)
  Heparan sulfate is one of the indicators of EG damage, and ANP & TNF-α, IL-6 are known to correlate with EG damage. So in this study, the investigators measure the plasma concentrations of Haparan sulfate, ANP & TNF-α, IL-6 as well as Syndecan-1, and also identify the overall short-term prognosis of the patients.
Composite rate of morbidity and mortality | If the hospitalization period is within 30 days, follow-up is done up to 30 days.
  Composite morbidity and mortality (Mortality, Stroke, Re-operation, Sternal infection, Prolonged ventilation, Renal dysfunction)
Composite rate of morbidity and mortality | If the hospitalization period exceeds 30 days, follow-up is done throughout the hospitalization period.
  Composite morbidity and mortality (Mortality, Stroke, Re-operation, Sternal infection, Prolonged ventilation, Renal dysfunction)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiac Anesthesiology, Department of Anesthesiology and Pain Medicine, Cardiovascular Hospital, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nan Z, Soh S, Shim JK, Kim HB, Yang YS, Kwak YL, Song JW. Effect of 5% albumin on endothelial glycocalyx degradation during off-pump coronary artery bypass. Can J Anaesth. 2024 Feb;71(2):244-253. doi: 10.1007/s12630-023-02652-7. Epub 2023 Nov 21. PMID 37989943